CLINICAL TRIAL: NCT07344142
Title: Improving Digital Wellbeing in Saudi Adolescents: Cluster-randomized Trial
Brief Title: Improving Digital Wellbeing in Saudi Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Aramco Services Company (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00023832
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Digital Technology Use; Social Media Addiction; Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): (1) treatment as usual (TAU) will receive the Ministry of Education (MOE) Digital Wellbeing Unit that is implemented in 12th grade as part of the Digital Citizenship Curriculum and a brief self-paced online teacher training
  Interventions: Behavioral: Digital Wellbeing Unit; Behavioral: Online Teacher Training
- Enhanced treatment (Experimental): (2) enhanced treatment including the MOE Digital Wellbeing Unit plus a WhatsApp-based intervention for parents and a brief self-paced online teacher training.
  Interventions: Behavioral: Digital Wellbeing Unit; Behavioral: Parent WhatsApp Groups; Behavioral: Online Teacher Training

INTERVENTIONS:
Behavioral: Digital Wellbeing Unit — (1) The student component utilizes the existing Digital Wellbeing Unit embedded within the national Digital Citizenship Curriculum, as implemented by the Saudi Ministry of Education. This curriculum is delivered by classroom teachers over the course of approximately one month, typically as part of standard instruction during the academic term. The content focuses on responsible digital media use, online safety, screen time awareness, and strategies for achieving digital balance. All instructional materials and delivery methods align with Ministry guidelines and are integrated into the regular school schedule.
Behavioral: Parent WhatsApp Groups — (2) The parental component, developed by the research team, is included in the enhanced intervention arm. It consists of structured engagement through WhatsApp groups formed with parents of students enrolled in the intervention schools. Parents in this group will receive daily messages for the duration of the curriculum delivery (approximately 4 weeks). These messages will include infographics, short expert video lectures, and brief videos designed to reinforce the concepts taught in the student curriculum. Content will focus on promoting healthy digital habits, improving communication between parents and children about technology use, and modeling appropriate digital behaviors at home.
  Arms: Enhanced treatment
Behavioral: Online Teacher Training — (3) Teachers in both arms will complete a brief self-paced online training (~45 minutes total) prior to delivering the Digital Wellbeing Unit. The training introduces key digital wellbeing concepts, provides implementation guidance aligned with the Ministry of Education curriculum, and includes resources to support classroom delivery. Completion will be monitored to ensure fidelity across schools.

SUMMARY:
Background: In Saudi Arabia, the rapid expansion of digital technology use-particularly among adolescents-has raised growing concerns about internet addiction and its impact on mental health and overall wellbeing. Building on formative work including national surveys, stakeholder interviews, and pilot testing, there is now a pressing need to rigorously evaluate interventions that can promote healthy digital habits among youth.

Study aims/objective: This study aims to evaluate the effectiveness of a school-based digital wellbeing intervention, with and without a supplemental parent engagement component, using a cluster randomized controlled trial design. The primary objective is to determine whether exposure to the student curriculum alone or in combination with a parent-focused intervention improves digital literacy, technology use behaviors, and psychosocial wellbeing among high school students. Secondary objectives include assessing changes in parent-child communication and parental attitudes toward digital media use.

Methods: Twenty (20) high schools across Qassim and Riyadh regions in Saudi Arabia will be randomly assigned to one of two study arms: (1) treatment as usual (TAU) will receive the Ministry of Education (MOE) Digital Wellbeing Unit that is implemented in 12th grad as part of the Digital Citizenship Curriculum and a brief self-paced online teacher training, or (2) enhanced treatment including the MOE Digital Wellbeing Unit plus a WhatsApp-based intervention for parents and a brief self-paced online teacher training. Approximately 125 students per school (~2,500 total) will complete surveys before and after the intervention period, assessing digital media habits, wellbeing, and communication patterns. Parent surveys will be administered in the enhanced arm to assess intervention engagement and parenting practices. Surveys with teachers will assess motivation and self-efficacy in delivering the digital wellbeing unit and fidelity of delivery.

Results: The study will generate evidence on the efficacy of school- and family-based strategies for improving adolescent digital wellbeing in the Saudi context. It will also provide insight into mechanisms of change, including the role of parental involvement in shaping adolescent digital habits.

Conclusion: Findings from this cluster randomized trial will inform national digital wellbeing policy and practice, offering a scalable model for youth-targeted behavioral health interventions in Saudi Arabia and similar settings.

ELIGIBILITY:
Inclusion Criteria:

* The study will include students enrolled in Grade 12 at participating high schools that are randomly assigned to one of the study arms.
* In addition, parents or legal guardians of these students will be eligible to participate in the parent-focused component of the intervention if the student is assigned to the enhanced curriculum group.

Exclusion Criteria:

* Students and parents will be excluded from the study if the students and parents do not provide assent or consent to participate, in accordance with ethical guidelines.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Weekday leisure screen-time hours assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Weekday (screen time for leisure)

SECONDARY OUTCOMES:
Social Media Disorder Scale | Baseline, pre-intervention, post-intervention (1 month)
  Social Media Disorder Scale: Score range from 9-45 with higher scores indicating higher degree of Social Media Disorder
Internet Gaming Disorder Scale-ShortForm (IGDS9-SF) | Baseline, pre-intervention, post-intervention (1 month)
  Internet Gaming Disorder Scale-ShortForm (IGDS9-SF): Score range from 9-45 with higher scores indicating higher degree of Internet Gaming Disorder
Digital wellbeing knowledge 1 assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Knowledge regarding digital wellbeing topics covered in the curriculum; items were developed by the research team: Score range from 0-10 with higher scores indicating more digital wellbeing knowledge
Digital well-being knowledge 2 assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Knowledge regarding digital wellbeing topics covered in the curriculum; items were developed by the research team: Score range from 3-15 with higher scores indicating more digital wellbeing knowledge
Digital well-being attitudes assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Attitudes regarding digital wellbeing topics covered in the curriculum; items were developed by the research team: Score range from 5-25 with higher scores indicating more favorable attitudes toward digital balance and healthy technology use
Digital well-being self-efficacy assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Self-efficacy regarding digital wellbeing topics covered in the curriculum; items were developed by the research team: Score range from 5-25 with higher scores indicating stronger digital wellbeing self-efficacy
Digital well-being behavior change 1 assessed by survey: notification-checking frequency | Baseline, pre-intervention, post-intervention (1 month)
  Self-reported changes in digital media habits or wellbeing practices as a result of the intervention; items were developed by the research team: This item captures unnecessary notification-checking frequency with score range 1-5 and higher scores indicating worse digital wellbeing behavior.
Digital well-being behavior change 2 assessed by survey: device use before sleep | Baseline, pre-intervention, post-intervention (1 month)
  Self-reported changes in digital media habits or wellbeing practices as a result of the intervention; items were developed by the research team: This item captures avoiding device use before sleep with score range 1-5 and higher scores indicating better digital wellbeing behavior.
Digital well-being behavior change 3 assessed by survey: engagement in non-digital activities | Baseline, pre-intervention, post-intervention (1 month)
  Self-reported changes in digital media habits or wellbeing practices as a result of the intervention; items were developed by the research team: This item captures engagement in non-digital activities with score range 1-5 and higher scores indicating better digital wellbeing behavior.
Digital well-being behavior change 4 assessed by survey: use of apps or tools to monitor and manage digital habits | Baseline, pre-intervention, post-intervention (1 month)
  Self-reported changes in digital media habits or wellbeing practices as a result of the intervention; items were developed by the research team: This item captures use of apps or tools to monitor and manage digital habits with score range 1-5 and higher scores indicating better digital wellbeing behavior.
Number of participants who upload phone screen shots of Screentime app | Baseline, pre-intervention, post-intervention (1 month)
  The investigators will explore feasibility of collecting objective data from students including screenshots of Screentime app
Weekend leisure screen-time hours assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Weekend day (screen time for leisure)
Weekday work/study screen-time hours assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Weekday (screen time for work/study)
Weekend work/study screen-time hours assessed by survey | Baseline, pre-intervention, post-intervention (1 month)
  Weekend day (screen time for work/study)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Thrul, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Supporting information will be shared upon reasonable request.
Access Criteria: Supporting information will be shared upon reasonable request.